CLINICAL TRIAL: NCT03304106
Title: Clinical Investigation of New CI Delivery Models in an Adult Nucleus CI Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAM 5417
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Sensorineural Hearing Loss, Bilateral; Cochlear Implant
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Newly Implanted CI Recipients (Experimental): Use of AI technology to assist in audiologist's evaluation and programming of new (standard of care-commercial) cochlear implant recipients
  Interventions: Device: Commercially available cochlear implant and AI system
- Existing CI recipients (Experimental): Use of AI technology to assist in audiologist's evaluation and programming of existing cochlear implant recipients
  Interventions: Device: Commercially available cochlear implant and AI system

INTERVENTIONS:
Device: Commercially available cochlear implant and AI system — Use of AI technology to assist in audiologist's evaluation and programming of cochlear implant recipients

SUMMARY:
Use of Artificial Intelligent (AI) technology to assist audiologists in programming cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

Newly implanted and existing recipient Groups (Groups 1 and 2):

* Age 12 and older
* Monosyllabic word score administered at 60dBA (2 lists) with an appropriately fit hearing aid in the ear to be implanted who are receiving a cochlear implant as standard of care
* Group 2: 3 months or greater combined experience with commercially available sound processors
* Fluent spoken English skills

Exclusion Criteria:

* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations
* Additional cognitive, medical or social handicaps that would prevent completion of all study requirements as determined by the Investigational team
* Unwillingness or inability of the subject to comply with all investigational requirements
* Use of an acoustic component in the implanted ear
* Less than 18 active electrodes
* Hybrid L Cochlear Implant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Midwest Ear Institute, Kansas City, Missouri
  - New York University, New York, New York
  - Hearts for Hearing, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cochlear Hearing Center Houston, Houston, Texas
  - Peak ENT Associates, Provo, Utah

REFERENCES:
- [Derived] Zwolan TA, Presley R, Chenier L, Buck B. Investigation of an Outcomes-Driven, Computer-Assisted Approach to CI Fitting in Newly Implanted Patients. Ear Hear. 2021 May/Jun;42(3):558-564. doi: 10.1097/AUD.0000000000000957. PMID 33027199

RESULTS

PARTICIPANT FLOW:
Groups:
- Newly Implanted CI Recipients: Newly implanted recipients
- Existing CI Recipients: Existing recipients
Period: Overall Study
Arm/Group | Newly Implanted CI Recipients | Existing CI Recipients
Started | 44 | 58
Completed | 31 | 56
Not Completed | 13 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Newly implanted recipients
- Group 2: Existing recipients
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 31 | 56 | 87
Age, Continuous [Mean (Full Range); unit: years] | 63.52 [23 to 90] | 56.98 [13 to 89] | 59.31 [13 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 16 | 34 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Hearing Loss [Mean (Full Range); unit: years] | 28.29 [3 to 56] | 28.39 [1 to 74] | 28.35 [1 to 74]
Duration of Device Use [Mean (Full Range); unit: months] | 0 [0 to 0] | 79.30 [1 to 305] | 51.04 [0 to 305]
Ear Tested [Number; unit: participants]
  Left | 15 | 29 | 44
  Right | 16 | 27 | 43
Type of Sound Processor [Count of Participants; unit: Participants] — Population: Group 1 participants had a newly implanted CI and Group 2 participants had an existing CI. Therefore the baseline measure of what Type of Sound Processor (exisiting) only applies to Group 2.
  Participants
    number analyzed (Participants) | 0 | 56 | 56
    Kanso | 0 | 1 | 1
    N6 | 0 | 49 | 49
    N7 | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Monosyllabic Word Recognition Scores (CNC) in Quiet
Description: Monosyllabic word recognition was scored in quiet using Consonant-Nucleus-Consonant (CNC) words. Scores are listed as percentage correct thus a higher score (percentage) means a better outcome.Group 1: Preoperative to postoperative percentage performance after 6 months of cochlear implant use. Group 2: Visit A to Visit B after 1 month of cochlear implant use.
Time Frame: Pre-operative/Visit A; Group 1: 6 months; Group 2: 1 month
Population: All participants with complete data set
Measure: Mean (Standard Deviation); unit: percentage of correct words
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 31 | 56
percentage of correct words
  Pre-operative/Visit A | 13.9 (15.2) | 60.1 (23)
  6-Month: number analyzed (Participants) | 31 | 0
  6-Month | 60.2 (17.2) |
  Visit B (1-Month): number analyzed (Participants) | 0 | 56
  Visit B (1-Month) |  | 59.1 (22)

ADVERSE EVENTS:
Time Frame: Time of enrollment through 6 months post-operatively (Group 1) and time of enrollment through 1 month follow-up (Group 2)
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/56
Serious Adverse Events (participants affected / at risk) | 5/31 | 1/56
Other Adverse Events (participants affected / at risk) | 17/31 | 6/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=31) | Group 2 (N=56)
Hospitalization secondary to losing consciousness from sinus bradycardia (Cardiac disorders) | 1 | 0
Hospitalization (General disorders) | 1 | 0
Parkinson's disease diagnosis (Nervous system disorders) | 1 | 0
Hospitalization for sepsis (Infections and infestations) | 1 | 0
Dizziness (Ear and labyrinth disorders) | 1 | 0
Vertigo and BPPV (Ear and labyrinth disorders) | 1 | 0
Abnormal heart rhythm requiring placement of pacemaker (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=31) | Group 2 (N=56)
Dizziness and imbalance (Ear and labyrinth disorders) | 1 | 0
Tongue numbness/mouth numbness (Injury, poisoning and procedural complications) | 1 | 0
Headaches (Nervous system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Change in taste (Injury, poisoning and procedural complications) | 1 | 0
Loss of hearing (Ear and labyrinth disorders) | 1 | 0
MAP too loud, unable to wear within 48hours of activation (Injury, poisoning and procedural complications) | 1 | 0
Swelling at CI site (Ear not specified) (Ear and labyrinth disorders) | 1 | 0
Altered taste post-op (Injury, poisoning and procedural complications) | 1 | 0
Occasional dizziness (Ear and labyrinth disorders) | 1 | 0
Sinus infection (Infections and infestations) | 1 | 0
Diffuse photodamage of the skin (Skin and subcutaneous tissue disorders) | 1 | 0
Jaw soreness (General disorders) | 1 | 0
Pain behind left ear (Ear and labyrinth disorders) | 1 | 0
Swelling in face and neck (Injury, poisoning and procedural complications) | 1 | 0
A window blind fell and hit head causing pain on head and neck (General disorders) | 1 | 0
Tinnitus began night of surgery after a window blind fell on head (Ear and labyrinth disorders) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Lip swelling (General disorders) | 1 | 0
Arthritis of carpometacarpal joint on left thumb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pinched nerve in back causing pain down right leg (Nervous system disorders) | 1 | 0
Left ear tinnitus following surgery (Injury, poisoning and procedural complications) | 1 | 0
Increased tinnitus (Ear and labyrinth disorders) | 1 | 0
Redness and swelling on implanted ear (Injury, poisoning and procedural complications) | 1 | 0
Intermittent dizziness (Ear and labyrinth disorders) | 1 | 0
Right ear pain (Ear and labyrinth disorders) | 1 | 0
Spitting suture at cochlear implant incision site (Injury, poisoning and procedural complications) | 1 | 0
Left facial pain (Nervous system disorders) | 1 | 0
Fatigue post-surgery (General disorders) | 1 | 0
Tingling, numbing and slight pain at coil/magnet site on head (Ear and labyrinth disorders) | 1 | 0
Patient experienced uncomfortable loudness (Injury, poisoning and procedural complications) | 0 | 1
Flinching to high frequency stimulation (Injury, poisoning and procedural complications) | 0 | 1
Loudness discomfort and increased tinnitus (Injury, poisoning and procedural complications) | 0 | 1
Right lower abdominal pain (General disorders) | 0 | 1
Hammer toe surgery left foot (Musculoskeletal and connective tissue disorders) | 0 | 1
MAP too loud; decreased speech perception in noise (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PIs, restricts sites from publishing site data or study data without sponsor review and approval.

DOCUMENTS (2):
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03304106/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT03304106/SAP_001.pdf